CLINICAL TRIAL: NCT00643812
Title: Improving Firearm Storage in Alaska Native Villages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Alaska Native Tribal Health Consortium (Other)
Responsible Party: David C. Grossman, MD, MPH, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-7504-E/G 03
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Suicide; Suicide, Attempted; Wounds and Injuries
Keywords: Firearm storage; Suicide; Unintentional injury; Alaska Native; Suicide Attempt
MeSH Terms: conditions — Suicide; Suicide, Attempted; Wounds and Injuries; Accidental Injuries | interventions — Family Characteristics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): The "Early" intervention arm received a gun locker at baseline
  Interventions: Other: Installation of gun locker in household
- 2 (Active Comparator): Households in this arm received a gun locker at 12 months following the baseline survey
  Interventions: Other: Installation of gun locker in household

INTERVENTIONS:
Other: Installation of gun locker in household — Households were randomized to 'early' and 'late' arms. Each household received a gun locker, which was installed in the household. Early arm received gun lockers at baseline.
  Other Names: Gun safes; Gun cabinets
  Arms: 1
Other: Installation of gun locker in household — Households were randomized to 'early' and 'late' arms. Each household received a gun locker, which was installed in the household. "Late" arm received the gun locker 12 months after baseline.
  Other Names: Gun safes; Gun cabinets
  Arms: 2

SUMMARY:
Rates of suicide among young Alaska Native males are over ten-fold higher than among a similar age cohort in the rest of the United States. A high proportion of these deaths are associated with firearms. Firearms are an important part of the subsistence lifestyle of this population, however restriction of access to guns by youth may be a promising strategy to reduce the risk of suicides in this population. Previous research conducted in the first phase of this project has demonstrated that about 75% of homes in rural southwest Alaskan villages have guns, and only about 15% of these guns are locked; 6% are loaded.

The aims of this specific phase of the study to execute a randomized trial of an intervention to improve firearm storage practices among residents of selected villages. Our hypothesis is that households receiving training and equipment to store firearms in gun lockers will be more likely to store their guns locked at 12 months, compared to households not receiving the intervention.

DETAILED DESCRIPTION:
Rates of suicide among young Alaska Native males are over ten-fold higher than among a similar age cohort in the rest of the United States. A high proportion of these deaths are associated with firearms. Firearms are an important part of the subsistence lifestyle of this population, however restriction of access to guns by youth may be a promising strategy to reduce the risk of suicides in this population. Recent work by the HIPRC has shown that locked guns are associated with a 73% reduced risk of suicide, compared to unlocked guns. Similar protective associations were found for unloaded guns. A recent pilot project to improve the storage of guns conducted in southwest Alaska increased the proportion of households having all guns locked from 15% to 85%. The aims of this proposed study are to estimate the prevalence of firearm ownership and of specific firearm storage practices among residents living in the Bristol Bay and Yukon-Kuskokwim regions of southwest Alaska and to work with the Alaska Native health corporations to plan and execute a randomized trial of an intervention to improve firearm storage practices among residents of selected villages. This 3-year study consists of two phases.

The first phase is a regional survey of households within 20 randomly selected villages in southwest Alaska to estimate the extent of firearm ownership and existing storage practices in these communities. This weighted sample would be extrapolated to an overall estimate of these variables for each of the two Native corporations in the region. The second phase of the study will be a two-arm randomized controlled trial of an intervention to increase the proportion of households that store all of their firearms in a locked safe. A secondary outcome will be to reduce the proportion of home reporting the presence of a loaded gun. Households will be randomly assigned to either an early or late intervention group. The 'early' intervention group will receive the intervention at baseline. The 'late' intervention group will receive the intervention 12 months after baseline. All eligible households within participating villages will be educated about the potential protective value of safe firearm storage practices, and then be offered a gun safe to store all of their firearms. Household adults will be trained to use the safe and to carefully restrict access to the guns by youth. Each household will complete a questionnaire about storage practices and important co-variates at baseline, 12 months, and 18 months. Data will be analyzed to detect differences, between groups, in the proportion of homes with unlocked guns, and loaded guns, at 12 and 18 months after baseline. We estimate that the enrollment of 350 homes at baseline should provide 90% power to detect differences of about 16-20 absolute percentage point difference between groups, depending on the baseline prevalence of these variables. This study has the potential to have an important effect on firearm storage patterns in a population at high risk for suicide. If proven successful, it could be disseminated throughout Alaska and other high risk communities.

ELIGIBILITY:
Inclusion Criteria:

* Households in six villages in Western Alaska that owned a gun, did not own a gun locker, adult age 21 or over

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2004-11; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Household firearm arm storage status: 1. Any unlocked guns in home; 2. Any loaded guns in home; 3. Any unlocked ammunition | 12 and 18 months after installation of the gun safe

CONTACTS AND LOCATIONS:
Overall Officials: David C GRossman, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Harborview Injury Prevention and Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Grossman DC, Stafford HA, Koepsell TD, Hill R, Retzer KD, Jones W. Improving firearm storage in Alaska native villages: a randomized trial of household gun cabinets. Am J Public Health. 2012 May;102 Suppl 2(Suppl 2):S291-7. doi: 10.2105/AJPH.2011.300421. Epub 2012 Mar 8. PMID 22401514